CLINICAL TRIAL: NCT03960372
Title: Using Information and Communication Technology in Public Education Activities to Promote Family Communication and Well-being in Hong Kong
Brief Title: Public Education to Promote Family Communication and Well-being
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The University of Hong Kong (Other)
Collaborators: The Hong Kong Jockey Club Charities Trust (Other)
Responsible Party: Sponsor
Other Study IDs: UW 19-247
Record Dates: First submitted 2019-05-02; First posted 2019-05-23 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2023-12

CONDITIONS: Family Relations
Keywords: Family

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: ICT activities — Public education activities using ICT to promote family communication, sharing happiness with family members, and well-being in the community.

SUMMARY:
With the increasing use of information and communication technology (ICT), family information can be easily accessed. Family information seeking was found to be associated with higher levels of family well-being. Alongside the growth in popularity of ICTs and its role in promoting family well-being, there is also a growing appreciation that ICTs such as internet-enabled devices and web-based applications can offer many advantages compared to traditional face-to-face approaches when delivering behaviour change programmes.

Given the increasing use of ICT and its potential advantages in public education, ICTs emerge as new strategies of high impact service delivery in different community public education activities, including community events and workshops. Although ICT use is common in daily practice, the application of ICT in implementing public education activities is not common, especially in activities that promote family well-being.

The SMART Family-Link Project is to use ICT in public education activities to promote family communication, sharing happiness with family members, and well-being in the community. The public education activities include community public education events and community public education workshops. The present study aims to assess participants' satisfaction toward the public education activities, the efficiency in activities implementation, and the effectiveness of public education activities. Feedback from participants will be collected by questionnaire survey and interviews. Participants' engagement and response will be observed by observers and video and/or photo-taking.

DETAILED DESCRIPTION:
The last few decades have seen a dramatic rise in the use of information and communications technology (ICT) and Internet access. According to the World Bank, 1.33 per cent of individuals in the world were using the Internet in 1996; in 2006, this figure rose to 17.58 %; by 2016, 45.91 % of individuals were using the Internet. Concurrently, there has been a dramatic rise in the number of mobile cellular subscriptions across the globe in the last two decades.

In line with the global trend, Hong Kong had 18.25 million mobile service subscribers in 2016. The Hong Kong Family and Health Information Trends Survey (FHinTs) under the FAMILY Project was conducted to monitor opinions and behaviours regarding family health, information use, and health communications. The investigator's results showed that ICT platforms such as online websites, social media, and instant messages are widely used in Hong Kong. In FHinTs 2016 survey, 82.6% of the respondents had smartphones, and 48.8% had tablets. Similar findings from the Nielsen Media Index 2017 year-end report showed that 97% of all internet users in Hong Kong were using smartphones to access the internet. The amount of time spent online each day was 3.2 hours and 94% of people aged 12 to 64 were using the internet.

With the increasing use of ICT, family information can be easily accessed. According to the findings from FHinTs 2016, ICT was increasingly used as a method of family information seeking: 66.7% of respondents sought family information from online websites, compared with 53.6% in 2009. About 30.9% sought family information from social media such as Facebook, and 22.8% sought family information from instant messaging platforms such as WhatApp. Family information such as recreation (46.6%), family heath (22.9%) and elderly-related topics (17.9%) were most commonly sought. Also, family information seeking was associated with higher levels of family health, happiness, harmony, and overall family well-being. The associations were observed regardless of the type of sharing methods, such as face-to-face sharing or sharing via ICT means.

Alongside the growth in popularity of ICTs and its role in promoting family well-being, there is also a growing appreciation that ICTs such as internet-enabled devices and web-based applications can offer many advantages compared to traditional face-to-face approaches when delivering behaviour change programmes. One of the biggest challenges that face-to-face intervention programmes face is diminishing reach and impact due to barriers to accessibility, cost-efficiency, flexibility to adapt to individuals, and structured intervention integrity. Using ICTs can address these barriers and may thus contribute to improving reach. ICT also helps facilitate access to interventions from a large variety of settings at all times, bringing the intervention to participants at times convenient to them and diminishing the influence of the situational constraints on intervention participation rates. The rise of ICT has created promising and potential new avenues and demand for implementing interventions related to mental health and parenting.

Given the increasing use of ICT and its potential advantages in public education, ICTs emerge as new strategies of high impact service delivery in different community public education activities, including community events and workshops.

The goal of the study is to evaluate participants' satisfaction to the activities and the effectiveness of ICT-related activities to enhance family communication, relationship and happiness.

A process evaluation will be performed to evaluate the process of each component of the program. Qualitative and quantitative assessments will be used to evaluate the effectiveness of the activities.

ELIGIBILITY:
Inclusion Criteria:

* Chinese-speaking
* Aged 18 years and above
* Able to complete the questionnaire

Exclusion Criteria:

* Subjects who fail to meet the inclusion criteria

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Social service users and general public
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2019-03-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Satisfaction to the community activities | Immediately after the activities
  Outcome-based questions will be used to assess the level of satisfaction toward the general performance of the community activities. The score for each question ranges from 1 to 5. The higher score indicates the higher satisfaction.

SECONDARY OUTCOMES:
Family communication time | Baseline and 1 month
  Outcome based question will be used to assess the communication time with family members. The score for each question ranges from 0 to 10. The higher score indicates the better outcome performance.
Family communication quality | Baseline and 1 month
  Outcome based questions will be used to assess the quality of communication with family members. The score for each question ranges from 1 to 5. The higher score indicates the better family communication quality.
Family relationship | Baseline and 1 month.
  Outcome based question will be used to assess the relationship with family members. The score for each question ranges from 0 to 10. The higher score indicates the better family relationship.
Family happiness | Baseline and 1 month
  Outcome based question will be used to assess the family happiness.The score for question ranges from 0 to 10. The higher score indicates the better in family happiness
Attitude and practice to share happiness with family and friends | Baseline, immediately after activities and 1 month
  Outcome based questions will be used to assess the attitude and practice on sharing happiness with family members and friends. The score for each question ranges from 0 to 10. The higher score indicates the better outcome performance

CONTACTS AND LOCATIONS:
Overall Officials: Tai-hing Lam, MD, Principal Investigator — The University of Hong Kong
Locations (1):
- The University of Hong Kong, Hong Kong, Hong Kong

REFERENCES:
- [Background] Breitenstein SM, Gross D, Christophersen R. Digital delivery methods of parenting training interventions: a systematic review. Worldviews Evid Based Nurs. 2014 Jun;11(3):168-76. doi: 10.1111/wvn.12040. Epub 2014 May 19. PMID 24842341
- [Background] Sanders MR, Baker S, Turner KM. A randomized controlled trial evaluating the efficacy of Triple P Online with parents of children with early-onset conduct problems. Behav Res Ther. 2012 Nov;50(11):675-84. doi: 10.1016/j.brat.2012.07.004. Epub 2012 Aug 18. PMID 22982082
- [Background] Zielinski JJ. [Duration of the disease and distribution of some clinical features in a group of epileptic outpatients]. Neurol Neurochir Pol. 1968 May-Jun;2(3):389-93. No abstract available. Polish. PMID 4972482
- [Derived] Sit SM, Lai AY, Kwok TO, Wong HW, Wong YL, Chow E, Kwok YK, Wang MP, Ho SY, Lam TH. Development and evaluation of two brief digital health promotion game booths utilizing augmented reality and motion detection to promote well-being at a gerontechnology summit in Hong Kong. Front Public Health. 2022 Sep 23;10:923271. doi: 10.3389/fpubh.2022.923271. eCollection 2022. PMID 36211703
- See also: The World Bank, 2016. Internet users (per 100 people). — http://data.worldbank.org/indicator/IT.NET.USER.P2?end=2014&start=1990